CLINICAL TRIAL: NCT04131803
Title: Efficacy and Safety of Probiotics Combined With Standard Chemotherapy Plus Targeted Therapy in Patients With Metastatic Colorectal Cancer: A Prospective, Open-Label，Randomized, Multi-center Clinical Trial
Brief Title: Probiotics Combined With Standard Chemotherapy Plus Targeted Therapy in Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other); Cancer Hospital of The University of Chinese Academy of Sciences (Unknown); Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DIFFERENCE
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2020-10

CONDITIONS: Unresectable Metastatic Colorectal Cancer
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bifico combined with chemotherapy plus targeted therapy (Experimental): Bifico combined with chemotherapy plus targeted therapy
  Interventions: Drug: Bifico combined with chemotherapy plus targeted therapy
- chemotherapy plus targeted therapy (Experimental): chemotherapy plus targeted therapy
  Interventions: Drug: chemotherapy plus targeted therapy

INTERVENTIONS:
Drug: Bifico combined with chemotherapy plus targeted therapy — Bifico combined with chemotherapy plus targeted therapy
  Other Names: Bifico+chemotherapy+targeted therapy
  Arms: Bifico combined with chemotherapy plus targeted therapy
Drug: chemotherapy plus targeted therapy — chemotherapy plus targeted therapy
  Other Names: chemotherapy+targeted therapy
  Arms: chemotherapy plus targeted therapy

SUMMARY:
Bifico (also known as "bifidobacterium trifidum live powder") is a probiotic preparation that has been marketed and widely used in China. The number of live bacteria of lactobacillus acidophilus and bifidobacterium per gram should not be less than 1.0×107CFU. At present, it is mainly used for diarrhea and abdominal distension caused by intestinal flora imbalance. It can also be used for treating mild to moderate acute diarrhea and chronic diarrhea. Lactobacillus acidophilus and bifidobacteria have been fully proved in basic studies to improve gut microbiological environment and inhibit colorectal cancer. A recent paper published by Nature Biomedical Engineering reported that chemotherapy can effectively enhance the efficacy of colon cancer by regulating intestinal flora. Based on the above evidence, we propose that the current standard chemotherapy plus targeted therapy regimen combined with Bifico can exert a more powerful synergistic anticancer effect. To sum up, this study put forward innovative joint regulating intestinal flora environment with standard chemotherapy and target therapy of new concept and mode, to assess Bifico combined with standard chemotherapy plus targeted therapy compared to standard chemotherapy plus targeted therapy for efficacy and safety of metastatic colorectal cancer, combined with the intestinal flora, probiotics patient blood DNA analysis, etc. New technology, explore flora index correlation with the prognosis of patients' immune system function, and its potential as a predictive marker. It is worth noting that this study will closely combine the current most advanced intestinal flora 16S microbial polymorphism detection and single-cell sequencing technology, so as to truly achieve accurate and individualized treatment, evaluation and prognosis prediction.

DETAILED DESCRIPTION:
Patients were randomized to either standard therapy (i.e., chemotherapy + targeted therapy) or standard therapy combined with Bifico. We will provide patients with first-line, second-line and third-line treatment with full intervention, including maintenance treatment. The standard treatment regimen, first-line (FOLFOX regimen + cetuximab) : oxaliplatin 85mg/m2 intravenous infusion 2 hours day1 + calcium leucofolate (LV) 400mg/m2 intravenous infusion 2 hours day1 + 5-fluorouracil (5-fu) 400mg/m2 intravenous infusion day 1, and then 1200mg/ (m2·day) ×2 days continuous intravenous infusion + cetuximab 500mg/m2 intravenous infusion over 2 hours day 1, repeat every 2 weeks. First-line treatment 4 to 6 months after the effective disease control or stable but still no radical surgery opportunity, can enter maintenance treatment: 5 - FU + LV (dose with a line), repeat every 2 weeks, or capecitabine oral 2 1250 mg/m2 / day day 1-14 + beacizumab 7.5 mg/kg intravenous day 1, repeat every 3 weeks, or stop the systemic treatment, until a progression, and immediately to the next line treatment; Second-line (FOLFIRI regimen + bevacizumab) : irinotegam 180 mg/m2 iv infusion over 30-90min day 1 + LV 400mg/m2 iv infusion 2 hours day 1 + 5-fu400 mg/m2 iv infusion day 1, then 1200mg/ (m2·day) ×2 days continuous intravenous infusion + bevacizumab 5mg/kg introvenious infusion day 1, repeat every 2 weeks. Third line: fuquinib 160mg oral 1/ day day 1-21, repeat every 28 days, or regofenil 5mg oral 1/ day day 1-21, repeat every 28 days. Bifico 2g oral 3/ day, take the medicine daily.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥18 years and ≤75 years
2. Histologically and radiologically confirmed colorectal adenocarcinomaImaging and/or pathology confirmed the presence of distal metastases
3. Multidisciplinary team (MDT) identifies unresectable metastatic colorectal cancer (mCRC)
4. RAS and BRAF genes are wild-type
5. The patient had no previous treatment for mCRC, including chemotherapy, surgery, radiotherapy, hepatic artery chemoembolization (TACE) and targeted therapy
6. Hematological function was normal (platelet > 90×109/L; White blood cell > 3×109/L; Neutrophil > 1.5×109/L)
7. Serum bilirubin ≤1.5 times the upper normal value (ULN), transaminase ≤5 times ULN
8. No ascites, normal coagulation function, albumin ≥35g/L
9. Child-push liver function was rated A
10. Serum creatinine is below the upper normal limit (ULN) or the calculated creatinine clearance rate of > 50ml/min (using Cockcroft-Gault formula)
11. ECOG score 2-0
12. Life expectancy > 3 months
13. Sign written informed consent
14. Willing and able to receive follow-up until death or study completion or study termination

Exclusion criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. Recurrence of primary tumor
2. Severe arterial embolism or ascites
3. A tendency to bleed or clotting disorder
4. Hypertensive crisis or hypertensive encephalopathy
5. Severe uncontrolled systemic complications such as infection or diabetes
6. Clinically serious cardiovascular diseases such as cerebrovascular accident (within 6 months before enrollment), myocardial infarction (within 6 months before enrollment), uncontrolled hypertension after appropriate drug treatment, unstable angina, congestive heart failure (nyha2-4), and arrhythmia requiring drug treatment
7. History of central nervous system disease (e.g. primary brain tumor, epilepsy beyond the control of standard treatment, any brain metastasis or stroke)
8. Other malignancies in the past 5 years (except basal cell carcinoma of skin and/or cervical carcinoma in situ after radical resection)
9. Received any drug under study or treatment with the same type of drug in the last 28 days before the study
10. Any residual toxicity from previous chemotherapy (except hair loss), such as peripheral neuropathy ≥NCI CTC v3.0 standard level 2
11. Is allergic to any of the drugs in the study
12. Pregnant and lactating women
13. Inability or unwillingness to comply with research protocols
14. The presence of any other disease, dysfunction due to metastatic lesions, or a suspected medical condition indicated a possible contraindication to the use of the study drug or a population at high risk for treatment-related complications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-11-25 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 1 year
  the proportion of patients with tumor size reduction of a predefined amount and for a minimum time period